CLINICAL TRIAL: NCT03044652
Title: Prospective, Open-label, Multicenter, Multinational, Randomized Trial to Investigate the Non-inferiority of Treatment With WO2085 Moisturising Cream in Comparison to a Cream With 0.1% Estriol in a Panel of Post-menopausal Women Suffering From the Symptoms of Vulvovaginal Dryness in a Parallel Group Design
Brief Title: Investigation of Non-inferiority of Treatment of Vulvovaginal Dryness With WO2085 Moisturising Cream in Comparison to a Cream With 0.1% Estriol
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dr. August Wolff GmbH & Co. KG Arzneimittel (Industry)
Collaborators: proDERM Institut für Angewandte Dermatologische Forschung GmbH (Unknown); Bremer Pharmacovigilance Service GmbH (Other); GCP-Service International Ltd. & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VFCr-12/2015; 2016-002199-28 (EudraCT Number)
Record Dates: First submitted 2016-12-21; First posted 2017-02-07 (Estimated); Last update posted 2017-07-14 (Actual); Status verified 2017-07

CONDITIONS: Vulvovaginal Atrophy
Keywords: Vulvovaginal Dryness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Medical Device: WO2085 Moisturising Cream (Experimental): WO2085 is a hormone-free Moisturizing Cream and is used to treat "vulvovaginal dryness" symptoms.
  Interventions: Device: WO2085 Moisturising Cream
- Drug: Estriol Cream 0.1% (Active Comparator): Estriol Cream 0.1% is a standard therapy for the treatment of vulvovaginal atrophy in postmenopausal women.
  Interventions: Drug: Estriol Cream 0.1%

INTERVENTIONS:
Device: WO2085 Moisturising Cream — 2.5 g of the investigational product WO2085 Moisturising Cream will be applied intravaginally, once daily in the evening. After improvement of the symptoms the frequency may be reduced by the patient as needed. In addition 0.5 g (1 fingertip unit) may be applied to the outer genital area as needed (also several times per day).
  Arms: Medical Device: WO2085 Moisturising Cream
Drug: Estriol Cream 0.1% — 0.5 g of the reference product Estriol Cream 0.1% will be applied intravaginally once daily in the evening for the first 3 weeks. Subsequently, the frequency will be reduced to twice a week for the last 3 weeks for all patients in this treatment group.
  Arms: Drug: Estriol Cream 0.1%

SUMMARY:
The aim of the study is to gain further experience with regard to the performance of the medical device WO2085 Moisturising Cream in comparison to a cream with 0.1% estriol.

DETAILED DESCRIPTION:
"Vaginal dryness" is defined as dryness, itching, burning and pain unrelated to sexual intercourse.

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal women with the subjective symptoms of "vulvovaginal dryness" with a sum score (0-16) of the parameters dryness, itching, burning and pain unrelated to sexual intercourse of at least 3 AND a VAS value "Overall impairment of daily life due to the condition "vulvovaginal dryness" > 0 on Visit 1.
* Last menstruation more than 12 months before Visit 1 OR bilateral oophorectomy with or without hysterectomy more than 3 months before Visit 1.
* Physical and mental healthy women as assessed by the medical history.
* PAP test performed within the last 12 months before Visit 1 and result less than PAP III.
* Signed written informed consent before participation in the Trial.
* Willingness to actively participate in the trial and to come to the scheduled visits.

Exclusion Criteria:

* Known hypersensitivity against any of the ingredients of the test products.
* Any indication in the medical history regarding an impairment of the hepatic, renal, gastrointestinal, cardiovascular, pulmonary, endocrinological or hematological system (especially venous and arterial thromboembolism, ischemic stroke, myocardial infarction, porphyria) if clinically relevant for this clinical trial (cf. contraindications and warnings for Estriol cream 0.1%).
* Known thrombophilic disorders (e.g. protein C, protein S or antithrombin deficiency).
* Breast cancer (acute and / or in the medical history or suspected).
* Estrogen-dependent tumor (acute and / or in the medical history or suspected, especially ovarian and / or endometrial carcinoma).
* Systemic hormonal replacement therapy (tablets, patches, injections, dermal products), or phytohormonal therapy or use of SERMs (inter alia anti-estrogens) within 3 months before Visit 1 and / or during the conduct of this trial.
* Intrauterine device (IUD) with progestogen (Mirena®, Jaydess®)
* Pathological findings in cancer screening (Papanicolaou III, III D - V in the cervical test)
* Pathological changes in the vaginal or cervix area, which are caused by estrogen deficiency (except symptoms and condition of "vulvovaginal dryness"), e.g. diminution of labia caused by estrogen deficiency, constricted introitus.
* Patients with known infectious diseases (e.g. hepatitis or HIV infection).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Total Severity Score of the Treatment of "vulvovaginal dryness" at 6 weeks. | Baseline, after 3 and 6 weeks
  "Vulvovaginal dryness" will be measured by the Total Severity Score. It is defined as the sum score of the single subjective symptom parameters dryness, itching, burning and pain unrelated to sexual intercourse, each scored from 0=none to 4=very severe. In total a range of 0=no complaints to 16=very severe complaints is possible. Differences to Baseline (Visit 1) of the Total Severity Score assessed after six weeks of treatment (Visit 3) serve as the primary endpoint for the test of non-inferiority.

SECONDARY OUTCOMES:
Overall impairment of daily life | 6 weeks
  Overall impairment of daily life due to the condition "vaginal dryness" (including subgroup analysis of patients with mild, moderate or severe impairment) will be measured by using a Visual Analogue Scale (VAS)
Global judgement of efficacy | 6 weeks
  The global judgement of efficacy will be assessed by the investigator and the patient according to the following scale: 1=very good to 4=poor.
Global judgement of tolerability | 6 weeks
  The global judgement of tolerability will be assessed by the investigator and the patient according to the following scale: 1=very good to 4=poor.
Adverse Events | after 3 and 6 weeks
  Adverse events will be documented on Visits after 3 and 6 weeks, respectively (and in the patient diary, if applicable).

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Christoph Abels, MD, PhD, Study Director — Dr. August Wolff GmbH & Co. KG Arzneimittel; Prof. Petra Stute, MD, PhD, Principal Investigator — Universitätsklinik für Frauenheilkunde, Inselspital Bern; Kirstin Deuble-Bente, MD, Principal Investigator — proDERM Institute for Applied Dermatological Research, Germany
Locations (5):
- Germany (4):
  - Dr. Gerick, Aachen
  - Praxis für die Frau, Mölln
  - proDERM Institute for Applied Dermatological Research, Schenefeld
  - Praxis für die Frau, Schwarzenbek
- Frauenklinik Inselspital Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bachmann G. Urogenital ageing: an old problem newly recognized. Maturitas. 1995 Dec;22 Suppl:S1-S5. doi: 10.1016/0378-5122(95)00956-6. PMID 8775770
- [Background] Biglia N, Peano E, Sgandurra P, Moggio G, Panuccio E, Migliardi M, Ravarino N, Ponzone R, Sismondi P. Low-dose vaginal estrogens or vaginal moisturizer in breast cancer survivors with urogenital atrophy: a preliminary study. Gynecol Endocrinol. 2010 Jun;26(6):404-12. doi: 10.3109/09513591003632258. PMID 20196634
- [Background] Stute P, May TW, Masur C, Schmidts-Winkler IM. Efficacy and safety of non-hormonal remedies for vaginal dryness: open, prospective, randomized trial. Climacteric. 2015;18(4):582-9. doi: 10.3109/13697137.2015.1036854. Epub 2015 May 22. PMID 25845406
- [Background] Management of symptomatic vulvovaginal atrophy: 2013 position statement of The North American Menopause Society. Menopause. 2013 Sep;20(9):888-902; quiz 903-4. doi: 10.1097/GME.0b013e3182a122c2. PMID 23985562